CLINICAL TRIAL: NCT05131607
Title: Prone to Supine Breast MRI Trial II, P2S2 MRI Trial
Brief Title: 21DIF039: Prone to Supine Breast MRI II, P2S2 Breast MRI Trial
Acronym: 21DIF039
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: CairnSurgical, Inc. (Industry)
Responsible Party: Principal Investigator, Roberta diFlorio-Alexander, Staff Physician, Radiology, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY02001039
Record Dates: First submitted 2021-10-15; First posted 2021-11-23 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supine MRI (Experimental)
  Interventions: Procedure: Supine MRI

INTERVENTIONS:
Procedure: Supine MRI — After completion of the standard prone MRI sequences the patient will be positioned supine, coils will be placed and baseline images will be obtained. Then a second dose of contrast equal to the first dose will be given, and additional images will be obtained
  Other Names: Prone to Supine Breast MRI II, P2S2 MRI Trial

SUMMARY:
The purpose of this study is to determine whether a supine breast MRI obtained with a second intravenous injection of gadolinium contrast immediately after a standard clinical prone breast MRI will provide sufficient tumor visualization to allow a Radiologist to define and outline the tumor edges ("segment" the tumor). Accurate segmentation will allow a 3-D image of the tumor to be generated to create a breast cancer locator (BCL) surgical device to in aid removal of breast cancers.

DETAILED DESCRIPTION:
The clinical pre-operative breast MRI exam will be obtained in the prone position with intravenous (IV) Gadolinium (Gd) contrast injection per standard of care clinical protocol. After completion of the standard clinical prone breast MRI, the participant will be re-positioned and the investigative supine breast MRI protocol with a second dose of IV Gd will be obtained. A second dose of contrast equal to the first dose will be given, and additional images will be obtained in the supine position. Subtraction images will be generated for both the prone and the supine sequences. It is hypothesized that the second contrast injection will generate tumor-to-fibroglandular contrast differences such that supine subtraction images will allow visualization and segmentation of the tumor equal to prone segmentation images. It is expected that the addition of a second injection of contrast will improve the ability to visualize and accurately segment the supine post-Gd images. While the total dose of gadolinium delivered in two injections is twice the amount normally given during a clinical prone breast MRI, this total dose is equal to that administered for other clinical MRI studies such as cardiac MRI.

No additional imaging or testing will be required for this research study following the standard clinical MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Female gender.
3. Histologic diagnosis of invasive breast cancer or ductal carcinoma in situ.
4. Tumor size at least 1 cm in diameter as visualized on mammogram or US.
5. A staging, pre-operative breast MRI is considered to be clinically indicated.
6. Ability to voluntarily provide informed consent to participate prior to any study-related assessments/procedures being conducted.

Exclusion Criteria:

1. Absolute contraindication to MRI, including presence of implanted electrical device. (pacemaker or neurostimulator incompatible with MRI), aneurysm clip, or metallic foreign body in or near eyes.
2. Severe claustrophobia.
3. Contraindication to the use of gadolinium-based intravenous contrast, including anaphylaxis. Any known history of nephrogenic systemic fibrosis (NSF).
4. History of median sternotomy.
5. Pregnancy. All women of child-bearing age will be questioned about possible pregnancy status. In women who are unsure of pregnancy status, a urine pregnancy test will be performed.
6. Patients who have received neoadjuvant chemotherapy for their current diagnosis.
7. Known compromised renal function including chronic, severe kidney disease (GFR < 30 ml/min/1.73m2), or acute kidney injury.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 45 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Difference in mean tumor-to-fibroglandular contrast ratio in prone compared to supine breast MRI | Day of standard clinical MRI, 1 day
  Determine the mean tumor-to-fibroglandular contrast in a two bolus intravenous contrast injection prone to supine breast MRI study and compare this to the mean tumor-to-fibroglandular contrast of a single-contrast injection prone to supine breast MRI study.

SECONDARY OUTCOMES:
Evaluate tumor visualization and segmentability on supine breast MRI exam with additional contrast injection obtained immediately after prone contrast breast MRI, and compare to tumor visualization and segmentability on clinical prone breast MRI. | Day of MRI, 1 day
  Compare the proportion of cases with successful agreement between radiologists' segmentation volumes in the double-contrast dose prone to supine MRI study to proportion of cases with successful agreement in the single-contrast dose prone to supine MRI using a Hausdorff Distance (HD) threshold < 1 cm.

OTHER OUTCOMES:
Evaluate time required for double contrast prone to supine exam compared to single contrast prone to supine exam. | Day of MRI, 1 day
  Determine the time required to obtain the double contrast prone to supine exam by recording start and stop times of both Supine and Prone MRI, using minutes and seconds. Compare exam time to single contrast prone to supine (prior study)

CONTACTS AND LOCATIONS:
Overall Officials: Roberta diFlorio-Alexander, MD, Principal Investigator — DHMC
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No